CLINICAL TRIAL: NCT02691195
Title: Ultrasound-guided Serratus Plane Block for the Quality of Recovery After Modified Radical Mastectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fujian Provincial Hospital (Other)
Responsible Party: Principal Investigator, Yao Yusheng, Associate professor, Fujian Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: K2016-1-07
Record Dates: First submitted 2016-02-15; First posted 2016-02-25 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Anesthesia
Keywords: Ultrasound; Serratus Plane Block; Quality of recovery
MeSH Terms: interventions — Ropivacaine; Anesthetics, Local; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- group control (Placebo Comparator): group control :Before induction of intravenous anesthesia, patients were received an ultrasound-guided serratus plane block, the serratus plane was injected with 0.9% Nacl 0.4ml/Kg.
  Interventions: Drug: 0.9% Nacl
- group SPB (Experimental): group SPB:Before induction of intravenous anesthesia, patients were received an ultrasound-guided serratus plane block, the serratus plane was injected with 0.5% ropivacaine 0.4ml/Kg.
  Interventions: Drug: Ropivacaine

INTERVENTIONS:
Drug: Ropivacaine — patients were received an ultrasound-guided serratus plane block, the serratus plane was injected with 0.5% ropivacaine 0.4ml/Kg.
  Other Names: local anesthetic
  Arms: group SPB
Drug: 0.9% Nacl — patients were received an ultrasound-guided serratus plane block, the serratus plane was injected with 0.9% Nacl 0.4ml/Kg.
  Other Names: Normal saline
  Arms: group control

SUMMARY:
Regional anesthesia improves quality of recovery after surgery in many studies. Ultrasound-guided serratus plane block is a novel technique which may be a viable alternative to current regional anesthetic techniques. This randomized, controlled trial is to examine the effects of ultrasound-guided serratus plane block anesthetic on the QoR after breast tumor resection.

DETAILED DESCRIPTION:
A total of 72 subjects (36 patients for each groups) were enrolled in this study. Patients were allocated to either the general anesthesia group (group control) or SPB (serratus plane block) + general anesthesia groups (group SPB) using randomized central computer-generated sequence software (SAS 19.0). The allocation ratio was 1:1 for the two groups. Group assignment was concealed by opaque sticking envelops. The major research content is to evaluate the quality of recovery using 40 questionnaire (QoR-40).

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists' (ASA) Physical Status class I-II scheduled for first modified radical mastectomy were included.

Exclusion Criteria:

* Patients with chronic ethanol
* long-term use of psychotropic drugs (e.g. sedative drugs and antidepressant);
* contraindications for serratus plane block including coagulopathy, infection at the puncture site;
* unable to cooperate with this research due to cognitive impairment, psychopathy or not willing for the hospital follow-up;
* administration of other test drugs or joining in other clinical study in 3 months before our study;
* received radiotherapy or chemotherapy before surgery;
* other conditions not allocated for this study out of the researchers' consideration.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2016-03-15 (Actual); Primary Completion 2017-06-12 (Actual); Study Completion 2017-06-14 (Actual)

PRIMARY OUTCOMES:
The quality of recovery | at 24 hours after surgery
  The primary outcome was the quality of recovery, which was assessed at 24 hours after surgery using a 40-item questionnaire (QoR-40).

SECONDARY OUTCOMES:
Postoperative pain intensity | at postoperative hours 0.5, 1, 2, 4, 8 and 24
  Postoperative pain intensity was rated at postoperative hours 0.5, 1, 2, 4, 8 and 24 with Visual Analogue Scale (VAS) ranging from 0 to 10, where 0 means no pain and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Yusheng Yao, PHD & MD, Principal Investigator — Fujian Provincial Hospital
Locations (1):
- Fujian Provincial Hospital, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blanco R, Parras T, McDonnell JG, Prats-Galino A. Serratus plane block: a novel ultrasound-guided thoracic wall nerve block. Anaesthesia. 2013 Nov;68(11):1107-13. doi: 10.1111/anae.12344. Epub 2013 Aug 7. PMID 23923989
- [Derived] Yao Y, Li J, Hu H, Xu T, Chen Y. Ultrasound-guided serratus plane block enhances pain relief and quality of recovery after breast cancer surgery: A randomised controlled trial. Eur J Anaesthesiol. 2019 Jun;36(6):436-441. doi: 10.1097/EJA.0000000000001004. PMID 31021882